CLINICAL TRIAL: NCT04647929
Title: Comparison of Surgical Treatment Options for Primary Congenital and Developmental Glaucomas
Acronym: STOP-Glaucoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding for the study could not be found.
Sponsor: University of Zurich (Other)
Collaborators: Johannes Gutenberg University Mainz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STOP Glaucoma
Record Dates: First submitted 2020-11-16; First posted 2020-12-01 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Primary Congenital Glaucoma; Developmental Glaucoma
Keywords: glaucoma; primary congenital glaucoma; developmental glaucoma
MeSH Terms: conditions — Hydrophthalmos; Glaucoma | interventions — Trabeculectomy

STUDY DESIGN:
Intervention Model Description: Te patients will be randomly assigned in a 1:1 ratio to either (1) Santen PRESERFLO implant (intervention arm) or (2) trabeculectomy (standard therapy) .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRESERFLO MicroShunt (Experimental): Patients will undergo Santen PRESERFLO MicroShunt implantation with intraoperative use of Mitomycin C 0.2mg/ml for 2 minutes.
  Interventions: Device: Santen PRESERFLO MicroShunt
- Trabeculectomy (Active Comparator): Patients will undergo trabeculectomy with intraoperative use of Mitomycin C 0.2mg/ml for 2 minutes.
  Interventions: Procedure: Trabeculectomy

INTERVENTIONS:
Device: Santen PRESERFLO MicroShunt — the PRESERFLO MicroShunt will be implanted to increase aqueous humor outflow
  Arms: PRESERFLO MicroShunt
Procedure: Trabeculectomy — a fornix-based trabeculectomy with a 3x4mm flap will be performed to increase aqueous humor outflow
  Arms: Trabeculectomy

SUMMARY:
Newborn and children can be affected by two subgroups of this disease: (1) primary congenital glaucoma (PCG) or (2) developmental glaucoma (DG). The primary aim of this study is to compare the Santen PRESERFLO implant to trabeculectomy in PCG and DG patients as second surgery after failed trabeculotomy or goniotomy.

DETAILED DESCRIPTION:
Glaucoma is a chronic, progressive disease, leading to blindness if untreated or insufficiently treated. It is characterized by a loss of optic nerve fiber and a glaucomatous optic disc excavation and, a corresponding pattern of visual field loss. Newborn and children can be affected by two subgroups of this disease: (1) primary congenital glaucoma (PCG) or (2) developmental glaucoma (DG). PCG and DG are treated surgically, either by goniotomy or by trabeculotomy as first approach, and not with topical hypotensive medications. Whenever these procedures have failed, the subsequent surgical procedure is usually trabeculectomy with Mitomycin C or the implantation of a glaucoma drainage device. However, there is a lack of evidence regarding the "optimal" surgical approach after failed goniotomy/trabeculotomy. Optimal treatment in this young group of patients with a long life expectancy is crucial to prevent blindness, allow them to participate in a "normal" school and work environment, and to minimize disease burdens for these patients and their families as well as to minimize costs for society. Consequently, there is the desire to find a procedure with a superior success rate and even fewer or less severe complications compared to trabeculectomy. Recently, the Santen PRESERFLO was introduced. The results proved fewer complications and comparable efficacy to trabeculectomy, according results presented at scientific meetings. Yet, there are no published studies to compare the both procedures. The primary aim of this study is to compare the Santen PRESERFLO implant to trabeculectomy in PCG and DG patients.

ELIGIBILITY:
Inclusion Criteria:

* Minors younger than 18 years of age with a diagnosis of Primary Congenital Glaucoma (PCG) or Developmental Glaucoma (DG) will be included
* participants must have had a failed trabeculotomy or goniotomy (once or twice) or one 360° trabeculotomy.

Exclusion Criteria:

* Individuals with eye pathologies other than glaucoma or, who underwent intraocular surgery within the last 6 months will not be included.
* patients who will not be willing to proceed with the entire follow-up of 6 months, or whose legal representative did not sign the informed consent will not be enrolled.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Efficacy 1 | at 6months compared to baseline (i.e. preop)
  Change in Goldmann-applanation intraocular pressure (IOP) in mmHg
Efficacy 2 | at 6months compared to baseline (i.e. preop)
  Change in the number of drug classes of intraocular pressure (IOP) lowering medications
Complication rate | within 6 months from surgery
  rate of intraoperative and postoperative complications (safety)

SECONDARY OUTCOMES:
Exome Sequencing | at baseline
  for known and susprected genes for primary congenital glaucoma or developmental glaucoma as a potential confounder for outcome and rates of complications will be statistically evaluated

CONTACTS AND LOCATIONS:
Overall Officials: - Individuals with eye pathologies other than glaucoma or, who Töteberg-Harms, MD, FEBO, Principal Investigator — University of Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Batlle JF, Fantes F, Riss I, Pinchuk L, Alburquerque R, Kato YP, Arrieta E, Peralta AC, Palmberg P, Parrish RK 2nd, Weber BA, Parel JM. Three-Year Follow-up of a Novel Aqueous Humor MicroShunt. J Glaucoma. 2016 Feb;25(2):e58-65. doi: 10.1097/IJG.0000000000000368. PMID 26766400
- [Result] Jayaram H, Scawn R, Pooley F, Chiang M, Bunce C, Strouthidis NG, Khaw PT, Papadopoulos M. Long-Term Outcomes of Trabeculectomy Augmented with Mitomycin C Undertaken within the First 2 Years of Life. Ophthalmology. 2015 Nov;122(11):2216-22. doi: 10.1016/j.ophtha.2015.07.028. Epub 2015 Aug 24. PMID 26315044